CLINICAL TRIAL: NCT02274376
Title: NIS Xeloda in Gastric Cancer
Brief Title: Non-Interventional Study of Xeloda (Capecitabine) in Patients With Gastric Cancer
Status: Completed | Type: Observational
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: ML21556
Record Dates: First submitted 2014-10-03; First posted 2014-10-24 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Cohort

SUMMARY:
This observational study will collect prospective data on the safety and tolerability of Xeloda in patients with advanced gastric cancer from every day clinical practice. Documentation of treatment for each patient is to continue until the end of treatment per oncologist's assessment.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged >/=18 years, with metastatic gastric cancer who are available for prospective documentation of their treatment (first-line chemotherapy)
* Informed consent

Exclusion Criteria:

* Contraindications to Xeloda per the Summary of Product Characteristics (SmPC)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with advanced gastric cancer eligible for Xeloda (capecitabine)
Sampling Method: Non-Probability Sample
Enrollment: 223 (Actual)
Dates: Start 2008-08; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Progression-free survival | Up to 4 years
Safety and tolerability: incidence and nature of adverse drug reactions | Up to 4 years

SECONDARY OUTCOMES:
Proportion of patients with modifications in Xeloda dosing | Up to 4 years
Average duration of treatment | Up to 4 years
Number of modifications in chosen regimen combination therapy | Up to 4 years
Incidence and nature of dose interruptions | Up to 4 years

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (1):
- Mannheim, Germany